CLINICAL TRIAL: NCT06190028
Title: Evaluation of Performance and Safety of IRIDIUM® A Gel Preservative-free Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension and Concomitant Dry Eye Syndrome on Multiple Long-term Topical Hypotensive Therapy: a Prospective, Multicentric, Open-label Clinical Investigation.
Brief Title: Evaluation of Performance and Safety of Carbopol 980 NF 0.2%- Based Medical Device in the Management of Patients With Glaucomar or Ocular Hypertension and Concomitant Dry Eye Syndrome on Multiple Long-term Topical Hypotensive Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS06-21-01
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye Syndrome; Glaucoma and Concomitant Dry Eye Syndrome; Ocular Hypertension and Concomitant Dry Eye Syndrome; Multiple Long-term Topical Hypotensive Therapy
MeSH Terms: conditions — Dry Eye Syndromes; Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IRIDIUM A gel (Experimental): Patients will receive IRIDIUM® A gel (four boxes to be used and one spare box) and they will be instructed to bilaterally apply 1 drop per eye onto the conjunctival sac 2 times a day for 60 days (one application during the day and one before going to sleep).
  Interventions: Device: Iridium A Gel

INTERVENTIONS:
Device: Iridium A Gel — IRIDIUM® A gel is a sterile, preservative free ophthalmic gel, containing Carbopol, amino acids, Echinacea and Aloe extract. IRIDIUM® A gel is indicated for the protection of the eye surface particularly at night, even in the presence of changes in histological continuity and blepharitic conditions, including those of an iatrogenic nature, following the use of hypotonic eye drops and of the preservatives contained therein.
  Other Names: Carbopol 0.2%

SUMMARY:
The main aim of this investigation is to evaluate the effect of the preservative-free ophthalmic solution IRIDIUM® A gel on the ocular surface of patients with glaucoma or OHT and concomitant DES under multiple long-term topical hypotensive therapy for at least 6 months. The underlying assumption is that ophthalmic solutions as adjuvants for the management of IOP- or glaucoma-associated dry eye may induce a protection of the eye surface with consequent improvement of the symptoms and of the overall quality of life.

DETAILED DESCRIPTION:
IRIDIUM® A gel is a sterile, preservative free ophthalmic gel, containing Carbopol, amino acids, Echinacea and Aloe extract. IRIDIUM® A gel is indicated for the protection of the eye surface particularly at night, even in the presence of changes in histological continuity and blepharitic conditions, including those of an iatrogenic nature, following the use of hypotonic eye drops and of the preservatives contained therein.

The main component of IRIDIUM® A gel is the Carbomer Carbopol 980 NF, a water-soluble polyacrylic acid with good mucoadhesion. It gives the gel the chemical-physical properties of viscosity and elasticity necessary for proper lubrication of the eyelids, forming a stable fluid film on the outer eye it provides protection to the eye surface, particularly at night.

The first approach to treat patients with ocular surface diseases relies on the use of artificial tears. Tear substitutes increase the volume of fluid on the ocular surface, thus reducing cell damage. Indeed, they induce a decrease in the osmotic pressure of the tear film and of the friction caused by eyelid movements.

For this, aqueous gels formulated using hydrophilic polymers along with those based on stimuli responsive polymers (in situ gelling or gel forming systems) continue to attract increasing interest for various eye health-related applications. Among these, eye drops containing carbomers or sodium hyaluronate are increasingly being used because of their non-Newtonian time-dependent response to shear strain, resulting in a longer ocular residence time.

Dry eye can also occur following specific treatments. In this regard, has been reported that dry eye symptoms are more prevalent in patients with IOP and/or glaucoma using topical IOP-lowering medications compared to the general population.

The evidence from literature suggests that different topical anti-IOP/glaucoma medications have different levels of impact on the health of the ocular surface. The main driver for this observation is the presence of preservatives in topical IOP-lowering medications. Generally, preservative-free medications have fewer adverse effects compared with preserved medications. However, the presence of preservatives, such as benzalkonium chloride (BAK), in antihypertensive eye drops used for long term therapy can cause ocular discomfort symptoms in glaucoma patients. BAK reduces the stability of the tear film by acting as a detergent on the lipid layer, by reducing the number of mucin secreting goblet cells, thus altering mucin presence and distribution over the ocular surface epithelium.

Clinicians need to take proactive decisions to manage ocular surface diseases of glaucoma patients as they are serious, chronic conditions. Previous findings confirm that glaucoma patients have a higher need for the use of artificial tears than age-matched controls , emphasizing that patients with ocular surface disease secondary to the chronic use of antiglaucoma medications should be preferably treated with preservative-free artificial tears.

ELIGIBILITY:
Inclusion Criteria:

1. Have an age ≥ 18 years,;
2. Have undergone the informed consent process and have signed an approved consent form;
3. Are able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and subjects able to cooperate with the Investigator and to comply with the requirements of the entire investigation (including ability to attend all the planned investigation visits according to the time limits), based on Investigator's judgement;
4. Have a diagnosis of glaucoma or Ocular Hypertension (OHT). Diagnosis of glaucoma will be based on: optic disc assessment, measurement of the retinal nerve fiber layer and neuroretinal rim with optical coherence tomography (OCT); characteristic repeatable visual field defects defined as a pattern standard deviation (PSD) with P < 0.05, and/or glaucoma hemifield test (GHT) results outside normal limits. Diagnosis of OHT will be based on history of IOP (intraocular pressure) > 21 mmHg in at least two occasions and normal optic disc and Humphrey visual field test;
5. Are receiving an ongoing topical therapy with two or more preserved ocular hypotensive agents (e.g. beta-blockers, alpha-agonists, carbonic anydhrase inhibitors, prostaglandins) for at least 6 months and are willing to continue these treatments at unchanged dose for the entire investigation duration;
6. Have a diagnosis of moderate to severe DES performed through the following exams: slit lamp examination (SLE), tear (lacrimal) meniscus exam, Schirmer's test, Tear Film Break-Up Time (TFBUT), fluorescein staining of the cornea and conjunctiva (Oxford Staining Scheme). Please note that a diagnosis of DES may be performed at entry in the investigation;
7. Have a Tear Film Break-Up Time (TFBUT) value < 7 sec;
8. Have performed a Humphrey Visual Field Test in the last 4 months, if not available the test will be performed during the screening visit;
9. In case of females of child-bearing potential (i.e., not permanently sterilized - post hysterectomy or tubal ligation status - or not postmenopausal), they must have a negative urine pregnancy test at T0 and use a reliable form of contraception for a least 1 month prior to T0 and throughout the investigation, according to the definition of Note 3 ofICH M3 Guideline*.

   * Note: According to the definition of Note 3 of ICH M3 Guideline a highly effective method is defined as those which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Highly effective birth control methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence.

Exclusion Criteria:

1. Best corrected visual acuity score < 20/40;
2. Ischemic oculopathy;
3. Contraindications to use of topical solution components used in this investigation or known allergy/hypersensitivity to any of the IRIDIUM®A gel ingredients;
4. Current use/use in the past 15 days of any ocular medications other than hypotensive eye drops;
5. Systemic treatments known to affect tear secretion;
6. Treatment with any other therapy that, according to Investigator's judgment, could interfere with the assessment of the efficacy or incidence of adverse events;
7. Any history or slit lamp evidence of eye surface diseases different from DES;
8. History of ocular trauma or surgery in the past 12 months;
9. History of cataract in the past 6 months;
10. Any history of corneal refractive surgery;
11. Use of systemic steroids or immunosuppressants;
12. Participation in another clinical study/investigation at the same time as the present investigation or within 30 days;
13. History of drug, medication or alcohol abuse or addiction;
14. Pregnant (positive urine pregnancy test) or breastfeeding women, or women planning to become pregnant during the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy Assessment of dry eye symptoms from baseline | Day 30
  Changes from baseline (T0) to Day 30 (T1) of the Impact of Dry Eye on Everyday Living (IDEEL) questionnaire ("Dry Eye Symptom-Bother" module) score following treatment with IRIDIUM® A gel. The "Dry Eye Symptom-Bother" module includes 20 items: Item 1 is scored on a 5-point Likert-like scale from 0 "none of the time" to 4 "all of the time"; Items 2-20 are scored on a 4-point Likert-like scale from 1 "not at all" to 4 "very much". Patients can also answer "I did not have this symptom / Not applicable" (scored 0).
Efficacy Assessment of vision-related function from baseline | Day 30
  Dry Eye Symptom-Bother" module includes 20 items: Item 1 is scored on a 5-point Likert-like scale from 0 "none of the time" to 4 "all of the time"; Items 2-20 are scored on a 4-point Likert-like scale from 1 "not at all" to 4 "very much". Patients can also answer "I did not have this symptom / Not applicable" (scored 0)

SECONDARY OUTCOMES:
Efficacy Assessment of dry eye symptoms from baseline | Day 60
  Change from baseline of the IDEEL questionnaire ("Dry Eye Symptom-Bother" module) score.
  The "Dry Eye Symptom-Bother" module includes 20 items: Item 1 is scored on a 5-point Likert-like scale from 0 "none of the time" to 4 "all of the time"; Items 2-20 are scored on a 4-point Likert-like scale from 1 "not at all" to 4 "very much". Patients can also answer "I did not have this symptom / Not applicable" (scored 0).
Efficacy assement of tear film stability | Day 30 and Day 60
  Change from baseline (T0) to Day 30 (T1) and Day 60 (T2) of the Tear Film Break-Up Time (TFBUT).
  This test is used to measure the tear film stability. Break-Up Time is defined as the time interval after a patient blink to the first appearance of dryness in the tear film. The patient is considered affected by dry eye if a dry area appears before 10 seconds
Changes on Intraocular pressure from baseline | Day 30 and Day 60
  IOP measurement, using Goldmann applanation tonometry. Tonometry is the technique used to determine the intraocular pressure (IOP), the fluid pressure inside the eye. Normal eye pressure ranges from 10 to 21 mmHg. Goldmann applanation tonometer is currently the most widely used device in clinical practice for IOP measurements and is considered criterionstandard due to its low cost, lack of consumables, simplicity, and integration into the workflow of the slit lamp examination in a busy clinic.
Assessment of patients' production of aqueous tears from baseline | Day 30 and Day 60
  Change from baseline the Schirmer's test I values. The Schirmer's test I is one of the commonly used methods to assess the aqueous tear production. A paper strip is inserted into the eye, under the eyelid, in the lower fornix near the lateral corner, away from the cornea, for five minutes to measure the production of tears. The wet portion of the strip is measured in millimeters. Values above 10 mm have to be considered normal
Assessment of ocular surface health from baseline | Day 30 and Day 60
  Change from baseline of the quality of the cornea and the conjunctiva, as measured using the Oxford Staining Scheme. Staining with fluorescein will be used to identify corneal and conjunctival epithelium defects. Indeed, the corneal surface will stain whenever there is a disruption of cell-to-cell junctions. The staining can show corneal superficial punctate epithelial erosions in patterns that are consistent with certain causes of dry eye
Assessment of conjunctival goblet cells (CGC) density and on the superficial corneal nerve fiber layer through confocal microscope | Day 30 and Day 60
  Confocal microscopy enables detailed investigation of tarsal and palpebral conjunctiva, central and peripheral cornea, tear film, and lids, and it allows evaluation of the ocular surface at the cellular level. The Heidelberg Retina Tomograph (HRT) is one of the well-established in vivo confocal imaging systems and, when combined with the "Rostock Cornea Module" (RCM), offers a new possibility for in vivo imaging histology for the visualization of the anterior segment of the eye.
  The parameters will be analysed manually or using automated measurements with image analysis software. For the Cornea, density of epithelial cells (number of cells), endothelial morphology (percentage of normal cells), density of endothelial cells (number of cells) will be assessed.
Assessment of conjunctival goblet cells (CGC) density and on the superficial corneal nerve fiber layer through confocal microscope | Day 30 and Day 60
  Confocal microscopy enables detailed investigation of tarsal and palpebral conjunctiva, central and peripheral cornea, tear film, and lids, and it allows evaluation of the ocular surface at the cellular level. The Heidelberg Retina Tomograph (HRT) is one of the well-established in vivo confocal imaging systems and, when combined with the "Rostock Cornea Module" (RCM), offers a new possibility for in vivo imaging histology for the visualization of the anterior segment of the eye.
  The parameters will be analysed manually or using automated measurements with image analysis software. For the Conjunctiva, morphology (percentage of normal cells), density of cells (number of cells) muciparous caliciform (goblet) cells (number of cells) will be assessed.
Assessment of conjunctival goblet cells (CGC) density and on the superficial corneal nerve fiber layer through confocal microscope | Day 30 and Day 60
  Confocal microscopy enables detailed investigation of tarsal and palpebral conjunctiva, central and peripheral cornea, tear film, and lids, and it allows evaluation of the ocular surface at the cellular level. The Heidelberg Retina Tomograph (HRT) is one of the well-established in vivo confocal imaging systems and, when combined with the "Rostock Cornea Module" (RCM), offers a new possibility for in vivo imaging histology for the visualization of the anterior segment of the eye.
  The parameters will be analysed manually or using automated measurements with image analysis software. For the fibre layer, fibre layer: number of nervous fibres, cells form (entire or fragmented cells) will be assessed.
Assessment of Incidence and nature of the Adverse Effects | Day 30 and Day 60
  Incidence and nature of the Serious Adverse Device Effects (SADEs); Incidence and nature of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs); Incidence and nature of the Adverse Device Effects (ADEs); Incidence and nature of Investigational Medical Device Deficiencies (IMDDs).

CONTACTS AND LOCATIONS:
Overall Officials: Michele Iester, MD, Principal Investigator — Ospedale Policlinico San Martino
Locations (3):
- Italy (3):
  - Policlinico San Martino, Genova
  - AOU Pisana Ospedale Cesanello, Pisa
  - IRCCS Fondazione G.B. Bietti, Roma

IPD SHARING:
Plan to Share IPD: No